CLINICAL TRIAL: NCT06627868
Title: Nicotinamide Adenine Dinucleotide (NAD+) Metabolism in Human Brown Adipose Tissue
Acronym: BATNAD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Responsible Party: Principal Investigator, Mueez U-Din, Adjunct Prof., University of Turku
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VARHA/13032/13.02.02/2024
Record Dates: First submitted 2024-10-02; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Obesity, Abdominal
MeSH Terms: conditions — Obesity, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- Oral NAD+ precursor supplementation (Experimental)
  Interventions: Dietary Supplement: NAD+ precursor

INTERVENTIONS:
Dietary Supplement: NAD+ precursor — NAD+ precursor supplementation (Nicotinamide, Nicotinamide Riboside, or Nicotinamide Mononucleotide)
  Arms: Oral NAD+ precursor supplementation
Other: Placebo — Oral placebo daily intake for 6 months
  Arms: Placebo

SUMMARY:
A fully functional brown fat helps maintain a healthy weight and decreases the risk of metabolic diseases such as type II diabetes (T2DM). Unfortunately, in human adults, the functionality of brown fat declines with age, and it is one of the reasons for gaining unhealthy weight, particularly around the waistline (central obesity). Currently, we do not clearly understand the reasons for the decline in brown fat functionality. It is possible that the decline in the availability of the molecule Nicotinamide Adenine Dinucleotide (NAD+), which is central to several metabolic processes, plays a role in the decline in brown fat metabolism. This project will clarify whether NAD+-based molecular-targeted therapies for the enhancement of whole-body insulin sensitivity and brown fat metabolism will be successful in adult humans, which will eventually be an important target for reducing the development of obesity and its comorbidities such as T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to provide informed consent to participate in the BATNAD study
* Must be able to read and speak English/Finnish/Swedish well enough to completely understand the instructions and provide informed consent
* Age 30-55 (sedentary lifestyle)
* BMI = 18-25 kg/m2 (normal-weight subjects)
* BMI ≥ 28 kg/m2 and waist circumference more than 100 cm in men and more than 90 cm in women (subjects with obesity)

Exclusion Criteria:

* Inability to have PET/CT (claustrophobia, metal implants, recent tattoo including metal components, weight > 200 kg)
* Pregnancy and pregnancy related conditions (postpartum/lactation during the last 12 months, or planning to become pregnant soon)
* Major alterations in the menstrual cycle (e.g., amenorrhea)
* Use of nicotine based products
* Hypo- or hyper- thyroidism (medical history, TSH, T3 or T4 levels out of the normal range)
* Diabetes mellitus (fasting Hb1Ac >6.5% or fasting glycaemia> 7.0 mmol/)
* Abnormal oral glucose tolerance test (2h OGTT > 11.1 mmol/L)
* Hypertension (blood pressure > 160/100 mmHg)
* Abnormal cardiovascular status (arrhythmia and/or long QTc in ECG, abnormal cardiac murmur, previous history of cardiovascular disease)
* Abnormal coagulopathy (e.g., clotting abnormality)
* Malignancies
* Immunological, autoimmune and primary/secondary immunodeficiency disorders (including or not any active treatment)
* Virus or bacterial infection (both asymptomatic and symptomatic picture) within the 45 days prior to the study start
* Vaccination within the 45 days prior to the study start
* Episode of fever or major surgery, burns and traumas within the month prior to the study start
* Chronic infections requiring chronic antibiotic or anti-viral treatment
* Whole blood donation in the last 3 months (>400 mL of blood) or plans for blood donation during the entire protocol period
* Weight change (intentional or not) over the last 6-months more than 5% of body weight, or plan to lose weight during the study
* Allergy to lidocaine or epinephrine, or other local anaesthetics
* Previous participation to studies where PET or CT method is used
* Use of any medication that, in the opinion of local clinician/researcher, would negatively impact or mitigate full participation and completion, or could influence the study results. This especially applies to the use of β or α adrenergic receptors agonists/antagonists (e.g., β-blockers).
* Any other cardiovascular, pulmonary, orthopaedic, neurologic, psychiatric or other conditions that, in the opinion of the local clinician/researcher, would preclude participation and successful completion of the protocol, or that would negatively impact or mitigate participation in and completion of the protocol

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-10-20 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Whole-body Insulin Sensitivity | 6 months
  Whole-body insulin sensitivity measured with hyperinsulinemic, euglycemic clamp technique

SECONDARY OUTCOMES:
Brown adipose tissue glucose uptake rate | 6 months
  Brown adipose tissue glucose uptake rate will be measured with 18F-FDG PET-CT imaging

CONTACTS AND LOCATIONS:
Overall Officials: Mueez U-Din, PhD, Principal Investigator — Turku PET Centre, Turku University Hospital; Kirsi A Virtanen, MD PhD, Principal Investigator — University of Turku
Locations (1):
- Turku PET Centre, Turku, Finland

IPD SHARING:
Plan to Share IPD: No